CLINICAL TRIAL: NCT02754544
Title: Pilot Investigation of Using Electrocorticogram (ECoG) in Predicting Eloquent Cortex and Post-Operative Functional Outcomes in Patients With Brain Tumors
Brief Title: Electrocorticography in Mapping Functional Brain Areas During Surgery in Patients With Brain Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-0775; NCI-2016-00794 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0775 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Brain Neoplasm; Metastatic Malignant Neoplasm in the Brain; Recurrent Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Masking Description: No Data Available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (electrocorticography) (Experimental): Patients undergo tumor resection. During surgery, patients also undergo electrocorticography with either the CorTec high resolution hybrid grid, the PMT high-resolution grid, or the Ad-Tech grid followed by direct electrocortical stimulation.
  Interventions: Procedure: Direct Electrocortical Stimulation; Other: Electrocorticography

INTERVENTIONS:
Procedure: Direct Electrocortical Stimulation — Undergo direct electrocortical stimulation
  Other Names: DCES; Direct Cortical Electrical Stimulation; Electrocortical Stimulation Mapping; ESM
Other: Electrocorticography — Undergo electrocorticography
  Other Names: ECoG

SUMMARY:
This pilot clinical trial studies how well electrocorticography works in mapping functional brain areas during surgery in patients with brain tumors. Using a larger than the standard mapping grid currently used during brain tumor surgery or a high-definition grid for electrocorticogram brain mapping may help doctors to better identify which areas of the brain are active during specific limb movement and speech during surgery in patients with brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To record electrocorticogram (ECoG) data intraoperatively with surface electrode grids during various motor, sensory (tactile) and speech tasks, and identify functional brain areas through the spectral analysis, and compare the preliminary data with our current pre-surgical mapping methods: functional magnetic resonance imaging (fMRI) and transcranial magnetic stimulation (TMS), and the gold standard, intraoperative direct electrical stimulation (DES).

SECONDARY OBJECTIVE:

I. To perform a preliminary assessment of the utility of using ECoG data in these patients to quantify new neurological and language/speech deficits in the short term (24 hours) and long-term (1, 3, and 6 months), and achieve a safe maximal tumor resection.

OUTLINE:

Patients undergo tumor resection. During surgery, patients also undergo electrocorticography with either the CorTec high resolution hybrid grid, the PMT high-resolution grid, or the Ad-Tech grid followed by direct electrocortical stimulation.

Following completion of study, patients are followed up within 24 hours from surgery and at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a tumor resection at the University of Texas M. D. Anderson Cancer Center for a newly diagnosed as well as recurrent primary or metastatic brain tumor located in or adjacent to motor and/or speech brain areas
* Patients >= 18 years of age
* Signed informed consent

Exclusion Criteria:

* Patients with significant neurological motor deficits of the upper extremities, and/or speech deficits, which would preclude them from performing the while awake intra-operative tasks at the discretion of the principal investigator (PI)
* Patients who have impaired vision and/or hearing and whose performance could affect the study will be excluded at the discretion of the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-07-22 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Electrocorticogram (ECoG) | Up to 6 months (± 4 weeks)
  Will be assessed by cortical electrical activity based on individual hand muscle function. ECoG will be compared to direct electrical stimulation (DES), navigated transcranial magnetic stimulation (nTMS), and functional magnetic resonance imaging (fMRI). The data obtained using ECoG will be correlated with the fMRI and TMS data acquired preoperatively and intraoperative DES. The categorical variables would be preoperative Karnofsky performance status and functional status, tumor location, fMRI, TMS, ECoG, and DES data points. Other variables involved in the analysis would be extent of resection and neurological and language/speech outcome. The Chi-square or Fisher's exact tests will be used to explore associations between categorical variables. Additional analysis may be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Sujit S Prabhu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org